CLINICAL TRIAL: NCT01586936
Title: Special Survey of Production of Antibody Against Coagulation
Brief Title: Non-Interventional Study of NovoSeven® Used as On-demand Treatment of Bleeds in Patients With Haemophilia A and B With Inhibitors
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7-1949
Record Dates: First submitted 2012-04-11; First posted 2012-04-27 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eptacog alpha users
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Prescription of eptacog alpha at the discretion of the physician

SUMMARY:
This study is conducted in Japan. The aim of this registry study is to observe the use of single dose and multi-dose use of eptacog alpha (NovoSeven®) and to compare short-term outcomes, including effectiveness, safety, quality of life and treatment satisfaction with the approved treatments.

ELIGIBILITY:
Inclusion Criteria:

* Treated with eptacog alpha (NovoSeven®)

Exclusion Criteria:

* Investigator decision to measure for antibody as unnecessary medical testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from general practice setting who have been deemed appropriate to receive NovoSeven® (eptacog alpha) as new treatment and as part of routine out-patient care by the prescribing physician
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 1999-03-10 (Actual); Primary Completion 2010-03-09 (Actual); Study Completion 2010-03-09 (Actual)

PRIMARY OUTCOMES:
Antibody production against eptacog alpha | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com